CLINICAL TRIAL: NCT02690714
Title: A Phase 2/3, Open-Label, Repeat-Dose Study of the Pharmacokinetics, Efficacy, and Safety of Prometic Plasminogen Intravenous Infusion in Subjects With Hypoplasminogenemia
Brief Title: A Study of Prometic Plasminogen IV Infusion in Subjects With Hypoplasminogenemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Prometic Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002C011G
Expanded Access: NCT03265171 (No longer available)
Record Dates: First submitted 2016-02-12; First posted 2016-02-24 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Hypoplasminogenemia; Congenital Plasminogen Deficiency
MeSH Terms: conditions — Congenital Plasminogen Deficiency | interventions — Plasminogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 6.6 mg/kg Plasminogen (Human) Intravenous (Experimental): 6.6 mg/kg Plasminogen (Human) Intravenous given every 2 to 4 days by a 10- to 30-minute intravenous infusion
  Interventions: Biological: Plasminogen (Human) intravenous

INTERVENTIONS:
Biological: Plasminogen (Human) intravenous — Prometic Plasminogen (Human) intravenous infusion given as single dose of 6.6 mg/kg in Segment 1 and repeat doses in Segments 2 and 3.

SUMMARY:
This is a Phase 2/3 pivotal study to evaluate pharmacokinetics (PK), efficacy, and safety of Prometic Plasminogen (Human) Intravenous Lyophilized Solution, the investigational medicinal product (IMP), in pediatric and adult subjects with hypoplasminogenemia.

DETAILED DESCRIPTION:
This is a Phase 2/3, open-label, repeat-dose study of the PK, efficacy, and safety of the IMP, in pediatric and adult subjects with hypoplasminogenemia. The study consists of a screening period and 3 treatment segments (Segment 1,2, and 3). Subjects who have documented individual PK profiles do not need to undergo Segment 1 and can proceed directly to Segment 2. Subjects in Segment 1 will receive a single dose of 6.6 mg/kg IMP infusion. Blood samples for PK analysis will be drawn prior to infusion and subsequently through 96 hours after the infusion to establish individual PK profiles. The sample drawn prior to infusion will be used to measure the subject's baseline anti-plasminogen antibody, plasminogen activity and antigen as well as D-dimer levels. The resulting PK profile will be used to determine each subject's dosing interval in Segment 2.

Based on individual PK profiles from Segment 1 subjects will receive 6.6 mg/kg IMP infusion every second, third, or fourth day for 12 weeks in Segment 2. For subjects who directly enter Segment 2, baseline assessments will be conducted before the first dose of IMP, including a blood sample to measure the baseline anti-plasminogen antibody, plasminogen activity and antigen as well as D-dimer levels. Subjects will visit the study sites on Week 1 and subsequently every 4 weeks, and receive the IMP infusion at the study site. Blood samples will be obtained at each study visit at Weeks 4, 8 and 12 and by a home health nurse at Weeks 2, 6 and 10. Subjects will undergo clinical assessments of the disease, including but not limited to: photographic measurements of visible lesions, spirometry for subjects with pulmonary involvement, and imaging study of nonvisible lesions, as applicable. Plasma samples will be drawn before IMP administration every 2 weeks to measure the trough levels of plasminogen activity and antigen, and D-dimer.

At the end of Segment 2, subjects will have the option to participate in Segment 3 where they will continue to receive IMP for an additional 36 weeks in Norway, and until product licensing or study termination by the sponsor for subjects in the United States. Subjects will return to the study sites for assessments every 3 months to monitor subjects' clinical status and plasminogen trough levels. Subjects at the Norway site in Segment 3 should return to the study site for a safety follow-up visit 30 days after the final IMP dose. Due to the delay in product approval, subjects at the US site in Segment 3 will be allowed to enroll in treatment protocol 2002C018G and continue ongoing IMP treatment without any break in treatment. If subjects decide to not enter treatment protocol 2002C018G, then they will stop IMP and return to the study site for a safety follow-up visit 30 days after the final IMP dose.

The primary objective of this study is to achieve an increase of individual trough plasminogen activity by at least an absolute 10% (i.e., 10 U/dL) from baseline during the 12 weeks of plasminogen replacement therapy in Segment 2; and to evaluate the efficacy of plasminogen replacement therapy on clinically evident or visible symptoms of hypoplasminogenemia during the 48 weeks of dosing in Segments 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or female between the ages of 2 and 80 years (inclusive), is able to provide informed consent or assent, and agrees to use contraceptive methods during the study (unless documented as biologically or surgically sterile or has not reached reproductive age).
* Subject has documented history of hypoplasminogenemia and has plasminogen activity level ≤ 45%.
* Subject had a documented history of lesions and symptoms consistent with a diagnosis of congenital plasminogen deficiency.
* Subject has documented vaccination to hepatitis A virus (HAV) and hepatitis B virus (HBV), or has received the first dose of HAV and HBV vaccine prior to the first dose of IMP and is scheduled to receive the second vaccine dose.

Exclusion Criteria:

* Subject has uncontrolled hypertension; clinical or laboratory evidence of an intercurrent infection; a malignancy within 3 years, except for basal or squamous cell skin cancer; a psychiatric disorder; chronic or acute clinically significant inter-current illness; or evidence of renal and hepatic dysfunction.
* Subject is pregnant or lactating
* Subject has a history of anaphylactic reactions to blood or blood products that may interfere with participation in study in the opinion of the investigator.
* Subject is a previous organ transplant recipient; has received exogenous plasminogen within 2 weeks of the screening; has a history of anaphylactic reactions to blood or blood products; or has received another IRB-approved interventional clinical trial of a drug, biologic, or device within 30 days before the first dose of the IMP.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2017-12-17 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Shapiro, MD, Principal Investigator — Indiana Hemophilia & Thrombosis Center
Locations (2):
- Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana, United States
- Oslo University Hospital HF, Oslo, Sognsvannvejen 20, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shapiro AD, Nakar C, Parker JM, Albert GR, Moran JE, Thibaudeau K, Thukral N, Hardesty BM, Laurin P, Sandset PM. Plasminogen replacement therapy for the treatment of children and adults with congenital plasminogen deficiency. Blood. 2018 Mar 22;131(12):1301-1310. doi: 10.1182/blood-2017-09-806729. Epub 2018 Jan 10. PMID 29321155
- [Derived] Shapiro AD, Nakar C, Parker JM, Thibaudeau K, Crea R, Sandset PM. Plasminogen, human-tvmh for the treatment of children and adults with plasminogen deficiency type 1. Haemophilia. 2023 Nov;29(6):1556-1564. doi: 10.1111/hae.14849. Epub 2023 Sep 6. PMID 37674358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 sites, 1 in the United States (US) and 1 in Norway. The first participant was screened in May 2016 and the last participant visit was in October 2018.
Groups:
- 6.6 mg/kg Plasminogen (Human) Intravenous: Prometic Plasminogen (Human) intravenous 6.6 mg/kg Plasminogen (Human) Intravenous given every 2 to 4 days by a 10- to 30-minute intravenous infusion for 48 weeks. Some subjects received more than 48 weeks of study drug.
Period: Segment 1: Single-dose Day -4 to Day 0
Arm/Group | 6.6 mg/kg Plasminogen (Human) Intravenous
Started | 9
Completed | 9 (Six participants skipped Segment 1 as they had PK data from Phase 1 study 2002C005G.)
Not Completed | 0
Period: Segment 2: Multi-dose Day 0 to Week 12
Arm/Group | 6.6 mg/kg Plasminogen (Human) Intravenous
Started | 15
Completed | 15
Not Completed | 0
Period: Segment 3: Extended Treatment Wks 12-48
Arm/Group | 6.6 mg/kg Plasminogen (Human) Intravenous
Started | 15
Completed | 15
Not Completed | 0
Period: Post-Wk 48: Safety Week 48 to EoS Visit
Arm/Group | 6.6 mg/kg Plasminogen (Human) Intravenous
Started | 12 (3 subjects from Norway did not go past 48 weeks)
Completed | 10
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | 6.6 mg/kg Plasminogen (Human) Intravenous
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.0 (13.05)
Age, Customized [Count of Participants; unit: Participants]
  2-11 years | 4
  12-17 years | 2
  > 17 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 1
  Non-Hispanic/Latino | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
  Norway | 3
Weight [Mean (Standard Deviation); unit: Kg] | 60.37 (26.803)
Visible and Non-Visible Lesions by Participant [Count of Participants; unit: Participants]
  None | 4
  >= 1 Visible or non-visible lesion | 11
Number of Visible and Assesable Non-Visible Lesions [Number; unit: Number of lesions]
  Number of lesions analyzed | 47
  Visible lesions | 32
  Non-visible lesions | 15
Plasminogen Activity [Mean (Standard Deviation); unit: % activity] — Plasminogen activity is a measurement of functional plasminogen levels. Plasminogen activity levels were measured with an automated chromogenic assay. Assay calibration curve was performed with a pool of normal human plasma with the assigned value of 100% plasminogen and plasminogen activity levels were reported in %. The normal reference range of plasminogen activity in healthy subjects was determined to be 70%-130% and the limit of quantification was set at 5%
  % activity | 21.1 (10.83)
Plasminogen Activity [Count of Participants; unit: Participants] — See note above
  Participants
    Plasminogen activity <5-10% | 3
    Plasminogen activity 11-20% | 4
    Plasminogen activity 21-30% | 6
    Plasminogen activity 31-40% | 1
    Plasminogen activity 41-45% | 1
    Plasminogen activity >45% | 0
Plasminogen antigen [Mean (Standard Deviation); unit: mg/dL] | 4.7 (3.7)
Plasminogen antigen [Count of Participants; unit: Participants]
  Plasminogen antigen <0.5-3.0 mg/dL | 4
  Plasminogen antigen 3.1-6.0 mg/dL | 10
  Plasminogen antigen 6.1-20.0 mg/dL | 1
  Plasminogen antigen >20.0 mg/dL | 0
Quality of Life Assessment [Count of Participants; unit: Participants] — For the QOL assessment, participants were asked to rate their overall QOL using a 11-point scale (0 =non-functioning, 10 = normal; The QOL scale was adapted from a scale developed by the American Chronic Pain Association.
  Participants
    QOL score = 0 | 0
    QOL score = 1 | 0
    QOL score = 2 | 0
    QOL score = 3 | 0
    QOL score = 4 | 0
    QOL score = 5 | 0
    QOL score = 6 | 1
    QOL score = 7 | 3
    QOL score = 8 | 1
    QOL score = 9 | 1
    QOL score = 10 | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Clinical Success in Number and Size of Lesions as Measured by Photographic or Other Imaging Modality Depending on the Organ System Affected or Change in Affected Organ Functionality at 48 Weeks.
Description: Overall clinical success was defined as 50% of participants with visible or other measurable lesions achieving at least a 50% improvement in lesion number/size or functionality impact from baseline. Visible lesions were defined as lesions that could be imaged and analyzed with digital photography. Non-visible lesions were defined as lesions whose dimensions could have been assessed by medical imaging studies (eg, computed tomography, magnetic resonance imaging, ultrasound, etc) or functional assessments (eg, spirometry, audiogram, oximetry, etc).Visible lesions that had both a length and width as measured by the 1mm scale, were referred to as "measurable lesions", and visible lesions that were too small to measure by the 1mm scale (length and/or width could not have been measured) were referred to as "non-measurable lesions".
Time Frame: 48 weeks
Population: Efficacy Population Week 48-Segment 3 included all 15 enrolled participants who completed the Week 48 visit at the time of the data cut-off date of 14Dec2017. This analysis included 11 participants with 47 visible and/or non-visible lesions at baseline. All 15 participants were assessed, however only 11 participants had visible and/or non-visible lesions at baseline.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 11
Number analyzed (Lesions) | 47
Lesions
  Total Visible/Non-Visible lesions resolved (%) | 34
  Total Visible/Non-Visible lesions improved (%) | 10
  Not applicable (not assessed) | 3

2. Primary Outcome: Number and Percentage of Particpants Who Achieved the Target Plasminogen Activity Trough Levels for at Least 3 Measurements in 12 Weeks During Segment 2
Description: Plasminogen activity is a measurement of functional plasminogen levels and is therefore the most accurate and specific method to quantify active Plasminogen (Human) Intravenous concentration in participants' plasma. Primary endpoint success was defined as at least 80% of evaluable participants (ie, 8 or more) achieving the target trough levels for at least 3 measurements in 12 weeks. The target trough level was defined as an increase in plasminogen activity level of at least an absolute 10% (10 U/dL) from the participant's individual baseline level.
Time Frame: 12 weeks
Population: Pharmacokinetic Population included any participant who had completed Segment 2 dosing and had provided at least 3 blood samples to measure plasminogen activity trough levels.
Measure: Count of Participants; unit: Participants
Groups:
- Plasminogen (Human) Intravenous: Prometic Plasminogen (Human) intravenous infusion given as single dose of 6.6 mg/kg in Segment 1 and repeat doses in Segment 2.
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 15
Participants | 15

3. Secondary Outcome: Overall Clinical Success in Number and Size of Lesions as Measured by Photographic or Other Imaging Modality Depending on the Organ System Affected or Change in Affected Organ Functionality at 12 Weeks
Description: as for outcome 1
Time Frame: 12 Weeks
Population: Efficacy population week 12 included all 15 enrolled participants who completed the week 12 visit. All 15 participants were assessed, however only 11 participants had visible and/or non-visible lesions at baseline.
Measure: Count of Units; unit: Number of Lesions
Units Other Than Participants: Number of Lesions
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 11
Number analyzed (Number of Lesions) | 47
Number of Lesions
  Total Visible/Non-Visible lesions resolved | 26
  Total Visible/Non-Visible lesions improved | 14
  Total Visible/Non-visible unchanged | 2
  Not applicable/Not assessed | 5

4. Secondary Outcome: Clinical Global Impression-Global Improvement (CGI-I) Scores at Week 12
Description: CGI-I scores are measured at 12 and 48 weeks after study drug treatment. The CGI-I Scale is a single, clinician completed scale designed to capture the clinician's impression of the participant's disease improvement over time.
  For this scale, clinicians were asked to consider their experience in this population and rate the change relative to the participant's state at Baseline using a 7-point scale (1 = very much improved, 7 = very much worse).
Time Frame: 12 weeks
Population: CGI-I population included all 15 enrolled participants who completed the week 12 (and week 48) visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 15
Participants
  CGI score 0 = Not assessed: Week 12 | 0
  CGI score 1 = Very much improved: Week 12 | 11
  CGI score 2 = Much improved : Week 12 | 4
  CGI score 3 = Minimally improved : Week 12 | 0
  CGI score 4= No change : Week 12 | 0
  CGI score 5 = Minimally worse : Week 12 | 0
  CGI score 6 = Much worse : Week 12 | 0
  CGI score 7 = Very much worse : Week 12 | 0

5. Secondary Outcome: Clinical Global Impression-Global Improvement (CGI-I) Scores at Week 48
Description: as for outcome 4
Time Frame: 48 Weeks
Population: CGI-I population included all 15 enrolled participants who completed the week 48 (and week 12) visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 15
Participants
  CGI Score 0= Not assessed: Week 48 | 0
  CGI Score 1= Very much improved: Week 48 | 13
  CGI Score 2= Much improved: Week 48 | 2
  CGI Score 3= Minimally improved: Week 48 | 0
  CGI Score 4= No change: Week 48 | 0
  CGI Score 5= Minimally worse: Week 48 | 0
  CGI Score 6= Much worse: Week 48 | 0
  CGI Score 7= Very much worse: Week 48 | 0

6. Secondary Outcome: Number of Participants With Improved Quality of Life (QOL) Score After 12 Weeks of Study Treatment
Description: Quality of life score (QOL) was measured at baseline and at 12 and 48 weeks after study drug treatment. For the QOL assessment, participants were asked to rate their overall QOL using an 11-point scale (0 = non-functioning, 10 = normal; The QOL scale was adapted from a scale developed by the American Chronic Pain Association.
Time Frame: 12 weeks
Population: Efficacy Population Week 48-Segment 3 included all 15 enrolled participants who completed the Week 48 visit at the time of the data cut-off date of 14Dec2017
Measure: Count of Participants; unit: Participants
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 15
Participants
  QOL score 0 : Week 12 | 0
  QOL score = 1 : Week 12 | 0
  QOL score = 2 : Week 12 | 0
  QOL score = 3 : Week 12 | 0
  QOL score = 4 : Week 12 | 0
  QOL score = 5 : Week 12 | 1
  QOL score = 6 : Week 12 | 0
  QOL score = 7 : Week 12 | 0
  QOL score = 8 : Week 12 | 0
  QOL score = 9 : Week 12 | 1
  QOL score = 10 : Week 12 | 13

7. Secondary Outcome: Number of Participants With Improved Quality of Life (QOL) Score After 48 Weeks of Study Treatment
Description: as for outcome 6
Time Frame: 48 weeks
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 15
Participants
  QOL Score 0: Week 48 | 0
  QOL Score 1: Week 48 | 0
  QOL Score 2: Week 48 | 0
  QOL Score 3: Week 48 | 0
  QOL Score 4: Week 48 | 0
  QOL Score 5: Week 48 | 1
  QOL Score 6: Week 48 | 0
  QOL Score 7: Week 48 | 0
  QOL Score 8: Week 48 | 0
  QOL Score 9: Week 48 | 1
  QOL Score 10: Week 48 | 13

8. Secondary Outcome: Plasminogen Activity Trough Levels Between Week 2 and Week 120
Description: Plasminogen activity trough levels were measured at Weeks 2, 4, 6, 8, 10, 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120.
Time Frame: Week 2 to Week 120
Population: Pharmacokinetic Population included any participant who had completed Segment 2, 3 and post week 48 dosing and had provided at least 3 blood samples to measure plasminogen activity trough levels.
Measure: Mean (Standard Deviation); unit: percentage of activity
Groups:
- Plasminogen (Human) Intravenous: Prometic Plasminogen (Human) intravenous infusion given as single dose of 6.6 mg/kg in Segment 1 and repeat doses in Segments 2,3 and post-week 48.
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 15
percentage of activity
  Week 2: number analyzed (Participants) | 14
  Week 2 | 45.1 (15.05)
  Week 4 | 48.9 (14.56)
  Week 6 | 52.4 (11.45)
  Week 8 | 48.3 (17.43)
  Week 10 | 50.2 (12.39)
  Week 12 | 51.0 (12.01)
  Week 24 | 45.0 (12.88)
  Week 36 | 45.5 (13.18)
  Week 48 | 41.7 (16.99)
  Week 60: number analyzed (Participants) | 13
  Week 60 | 49.0 (8.88)
  Week 72: number analyzed (Participants) | 12
  Week 72 | 46.7 (10.97)
  Week 84: number analyzed (Participants) | 12
  Week 84 | 51.7 (20.76)
  Week 96: number analyzed (Participants) | 9
  Week 96 | 50.1 (20.08)
  Week 108: number analyzed (Participants) | 7
  Week 108 | 45.0 (25.19)
  Week 120: number analyzed (Participants) | 2
  Week 120 | 36.5 (12.02)

9. Secondary Outcome: Plasminogen Antigen Trough Levels Between Week 2 and Week 120
Description: Plasminogen antigen trough levels were measured at Weeks 2, 4, 6, 8, 10, 12, 24, 36, 48, 60, 72, 84, 96, 108, and 120.
Time Frame: Week 2 to Week 120
Population: Pharmacokinetic Population included any participant who had completed Segment 2, 3 and post week 48 dosing and had provided at least 3 blood samples to measure plasminogen antigen trough levels.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Plasminogen (Human) Intravenous: Prometic Plasminogen (Human) intravenous infusion given as single dose of 6.6 mg/kg in Segment 1 and repeat doses in Segments 2, 3 and post-week 48.
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 15
mg/dL
  Week 2: number analyzed (Participants) | 14
  Week 2 | 6.550 (3.0457)
  Week 4 | 7.800 (3.8813)
  Week 6 | 7.268 (3.3155)
  Week 8 | 6.607 (3.0046)
  Week 10 | 9.460 (7.1543)
  Week 12 | 7.340 (2.9342)
  Week 24 | 5.913 (2.2181)
  Week 36 | 6.667 (2.7336)
  Week 48 | 6.973 (3.1299)
  Week 60: number analyzed (Participants) | 13
  Week 60 | 6.415 (1.7578)
  Week 72: number analyzed (Participants) | 12
  Week 72 | 6.083 (2.2851)
  Week 84: number analyzed (Participants) | 12
  Week 84 | 7.183 (3.8129)
  Week 96: number analyzed (Participants) | 9
  Week 96 | 7.656 (4.2030)
  Week 108: number analyzed (Participants) | 7
  Week 108 | 6.529 (4.0852)
  Week 120: number analyzed (Participants) | 2
  Week 120 | 6.550 (6.2933)

10. Secondary Outcome: Half-life (t1/2) of Plasminogen Activity After First Dose and at Week 12
Description: t1/2 is time required for the plasma concentration of Plasminogen to decrease 50% in the final stage of its elimination
Time Frame: First dose and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 15
Hours
  Mean (SD) t1/2 of plasminogen after the first dose | 34 (11.73)
  Mean (SD) t1/2 of plasminogen at week 12 | 39.2 (6.22)

11. Secondary Outcome: AUClast of Plasminogen Activity After the First Dose and at Week 12
Description: AUCLast is the area under the plasma concentration-curve of Plasminogen from time 0 to the last measured concentration.
Time Frame: First dose and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr*%
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 15
hr*%
  Mean (SD) AUClast after first dose of plasminogen | 3063.6 (778.67)
  Mean (SD) AUClast at Week 12 | 4656.0 (1012.66)

12. Secondary Outcome: Cmax of Plasminogen Activity After First Dose and at Week 12
Description: Cmax is the maximum plasma concentration of Plasminogen
Time Frame: First dose and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % plasminogen activity
Groups:
- Plasminogen (Human) Intravenous: Prometic Plasminogen (Human) intravenous Plasminogen (Human) intravenous: Prometic Plasminogen (Human) intravenous infusion given as single dose of 6.6 mg/kg in Segment 1 and repeat doses in Segment 2.
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 15
% plasminogen activity
  Mean (SD) Cmax of plasminogen after first dose | 95 (23.5)
  Mean (SD) Cmax of plasminogen at Week 12 | 125 (23.3)

13. Secondary Outcome: Cl of Plasminogen Activity After First Dose and at Week 12
Description: Cl is the volume of plasma cleared of Plasminogen per unit time
Time Frame: First dose and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 15
mL/hr/kg
  Mean (SD) Cl of plasminogen after first dose | 1.44 (0.460)
  Mean (SD) Cl of plasminogen at Week 12 | 0.92 (0.257)

14. Secondary Outcome: AUCinf of Plasminogen Activity After First Dose and at Week 12
Description: AUCinf is the area under the plasma concentration-curve of Plasminogen from time 0 extrapolated to infinity
Time Frame: First dose and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr*%
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 15
hr*%
  Mean (SD) AUCinf of plasminogen after first dose | 3605.8 (1023.88)
  Mean (SD) AUCinf of plasminogen at Week 12 | 5731.8 (1431.70)

15. Secondary Outcome: MRTlast for Plasminogen Activity After First Dose and at Week 12
Description: MRTLast is the mean residence time of Plasminogen from time 0 to the last measured concentration
Time Frame: First dose and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 15
hours
  Mean (SD) MRTlast of plasminogen after first dose | 30.6 (3.22)
  Mean (SD) MRTlast of plasminogen at Week 12 | 33.5 (1.60)

16. Secondary Outcome: Vss for Plasminogen Activity After First Dose and at Week 12
Description: Vss is the apparent volume of distribution at steady state of Plasminogen
Time Frame: First dose and 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Plasminogen (Human) Intravenous
Number analyzed (Participants) | 15
mL/kg
  Mean (SD) Vss of plasminogen after first dose | 63.3 (11.44)
  Mean (SD) Vss of plasminogen at Week 12 | 49.3 (10.36)

ADVERSE EVENTS:
Time Frame: Safety was assessed during the treatment period (up to 124 weeks) and a 30-day post-treatment period.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study drug treatment.
Groups:
- 6.6 mg/kg Plasminogen (Human) Intravenous: 6.6 mg/kg Plasminogen (Human) Intravenous given every 2 to 4 days by a 10- to 30-minute intravenous infusion for 48 weeks (Norway) and longer until product licensing or study termination by the Sponsor (US).
  Plasminogen (Human) intravenous: Prometic Plasminogen (Human) intravenous infusion given as single dose of 6.6 mg/kg in Segment 1 and repeat doses in Segments 2 and 3.
Arm/Group | 6.6 mg/kg Plasminogen (Human) Intravenous
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 6.6 mg/kg Plasminogen (Human) Intravenous (N=15)
Ileus (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Ear operation (Surgical and medical procedures) | 1
Ossiculoplasty (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 6.6 mg/kg Plasminogen (Human) Intravenous (N=15)
Lymph node pain (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Cardiac flutter (Cardiac disorders) | 1
Ehlers-Danlos syndrome (Congenital, familial and genetic disorders) | 1
Deafness unilateral (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Excessive cerumen production (Ear and labyrinth disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Motion sickness (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1
Conjunctival deposit (Eye disorders) | 1
Eye discharge (Eye disorders) | 2
Eye inflammation (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain lower (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 6
Aphthous ulcer (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Crohn's disease (Gastrointestinal disorders) | 1
Dental carries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
Gastric dilatation (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Paraesthesia oral (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Tooth development disorder (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 2
Chest discomfort (General disorders) | 2
Chills (General disorders) | 1
Fatigue (General disorders) | 3
Feeling abnormal (General disorders) | 1
Influenza like illness (General disorders) | 2
Infusion site bruising (General disorders) | 1
Infusion site discomfort (General disorders) | 1
Infusion site erythema † (General disorders) | 2
Infusion site extravasation (General disorders) | 4
Infusion site pain (General disorders) | 4
Infusion site rash (General disorders) | 1
Infusion site swelling (General disorders) | 4
Pain (General disorders) | 1
Peripheral swelling (General disorders) | 2
Pyrexia (General disorders) | 6
Seasonal allergies (Immune system disorders) | 2
Bronchitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 3
Fungal infection (Infections and infestations) | 1
Gastroenteritis norovirus (Infections and infestations) | 1
H1N1 influenza (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 10
Pharyngitis streptococcal (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 4
Tonsilitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Viral upper respiratory tract infection (Infections and infestations) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 2
Procedural vomiting (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2
Scratch (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Tongue injury (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 1
Blood iron decrease (Investigations) | 1
Blood pressure systolic increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Progesterone decreased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Burning sensation (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 8
Migraine (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Post-traumatic headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 2
Ovulation pain (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Uterine pain (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2
Vulvovaginal pain (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Oropahryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 3
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 2
Tumour pruritis (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Artificial crown procedure (Surgical and medical procedures) | 1
Central venous catheter removal (Surgical and medical procedures) | 1
Tooth repair (Surgical and medical procedures) | 1
Venipuncture (Surgical and medical procedures) | 1
Wisdom teeth removal (Surgical and medical procedures) | 1
Flushing (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 2
Dystension (Vascular disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of data generated in the study is governed by the Investigator Clinical Trial Agreement

DOCUMENTS (2):
  • Study Protocol (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT02690714/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT02690714/SAP_001.pdf